CLINICAL TRIAL: NCT02132390
Title: Study of Adjuvant Toremifene With or Without Goserrelin in Premenopausal Women With Stage I-IIIA, Hormonal Receptor Positive Breast Cancer Accompanied With or Without Chemotherapy Induced Amenorrhoea
Brief Title: Adjuvant Toremifene With or Without Goserrelin in Premenopausal Women With Stage I-IIIA, Hormonal Receptor Positive Breast Cancer Accompanied With or Without Chemotherapy Induced Amenorrhoea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, ZHOU Yidong, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUMCH-Breast-CIA
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer; Chemotherapy Induced Amenorrhea; Ovarian Function Suppression
Keywords: Breast cancer; Chemotherapy induced amenorrhea; Goserelin
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Toremifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients who didn't have CIA receive oral toremifene daily. Treatment continues for 5 years in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Toremifene
- Arm II (Experimental): Patients who had CIA receive toremifene as in arm I
  Interventions: Drug: Toremifene
- Arm III (Experimental): Patients without CIA receive oral toremifene and goserelin for ovarian function suppression
  Interventions: Drug: Goserelin
- Arm IV (Experimental): Patients with CIA receive oral toremifene and goserelin for ovarian function suppression.
  Interventions: Drug: Goserelin

INTERVENTIONS:
Drug: Goserelin
  Other Names: Zoladex
  Arms: Arm III; Arm IV
Drug: Toremifene
  Arms: Arm I; Arm II

SUMMARY:
Compare the potential benefits of adjuvant toremifene with or without goserelin in premenopausal women with stage I-IIIA, hormonal receptor positive breast cancer accompanied with or without chemotherapy induced amenorrhoea.

DETAILED DESCRIPTION:
This is a single center, randomized, controlled study. Patients undergo surgical resection with standard Doxorubicin/Cyclophosphamide Followed by Docetaxel (AC-T).

Chemotherapy begins within 4 weeks after surgery for patients randomized to arm I-IV. Arm I: patients who didn't have CIA receive oral toremifene daily. Treatment continues for 5 years in the absence of disease progression or unacceptable toxicity. Arm II: patients who had CIA receive toremifene as in arm I. Arm III: patients without CIA receive oral toremifene and goserelin for ovarian function suppression. Arm IV: patients with CIA receive oral toremifene and goserelin for ovarian function suppression. Patients are followed every 6 months for 5 years and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures
* Age of at least 18 and at most 45 years
* Spontaneous and regular menstrual periods before study entry with FSH below 15 mlU/ml in follicular phase
* Histologically confirmed primary breast cancer with the need for anthracycline-based chemotherapy
* Steroid receptor (estrogen and progesterone) positive tumor (diagnosis according to hospital standard-procedures)
* No clinical evidence of local recurrence or distant metastases. Complete staging work-up within 3 months prior to registration. All patients must have (bilateral) mammography or breast MRI, chest X-ray; other tests may be performed as clinically indicated
* Karnofsky-Index >80%
* Life expectancy of at least 10 years, disregarding the diagnosis of cancer
* Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution
* Patients underwent standard Doxorubicin/Cyclophosphamide Followed by Docetaxel (AC-T)
* Patients must be available for and compliant to treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compounds or incorporated substances
* Prior cytotoxic treatment for any reason
* Suspected (primary or secondary) ovarian insufficiency
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration and must implement adequate non-hormonal contraceptive measures during study treatment; prior use of hormonal contraceptives has to be discontinued before first Goserelin injection
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix)
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy
* Concurrent treatment with sex hormones. Prior treatment must be stopped before study entry

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-05; Primary Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | up to 120 months
Overall Survival | up to 120 months

SECONDARY OUTCOMES:
Quality of life | up to 120 months
Bone mineral density loss | up to 120 months
  measured by dual energy X-ray absorptiometry scans at every 12 months and by serum biomarkers
Hormone levels | up to 120 months
Incidence of pregnancy | up to 120 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China